CLINICAL TRIAL: NCT01834209
Title: Open-Label Study of Abiraterone Acetate Plus Prednisone in Asymptomatic or Mildly Symptomatic Subjects With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of Abiraterone Acetate Plus Prednisone in Asymptomatic or Mildly Symptomatic Patients With Metastatic Castration-Resistant Prostate Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100946; 212082PCR3012 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-04-15; First posted 2013-04-17 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Prostate Neoplasms
Keywords: Prostate neoplasms; Prostate cancer; Metastatic prostate cancer; Metatatic castration resistant prostate cancer; Abiraterone acetate; Prednisone; Prednisolone; Early access program
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; Prednisolone

INTERVENTIONS:
Drug: Abiraterone acetate — Abiraterone 1000 mg (4 x 250 mg tablets) taken orally once daily for 28-day cycles
Drug: Prednisone or prednisolone — 5 mg tablet taken orally once daily

SUMMARY:
The purpose of this study is to collect additional safety data during treatment with abiraterone acetate plus prednisone or prednisolone among adult participants with asymptomatic or mildly symptomatic metastatic castration-resistant prostate cancer (mCRPC) who reside in areas in which abiraterone acetate is not yet available for this indication through local healthcare providers, and who are not eligible for enrollment into an available ongoing clinical study of abiraterone acetate.

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known) early access protocol (EAP). Approximately 60 participants will be enrolled in this study. Participants will receive abiraterone acetate 1000 mg daily plus prednisone or prednisolone 5 mg daily. Treatment in 28-day cycles will continue until progression of clinical disease. Study drug will be provided until the company obtains market authorization and reimbursement in the participant countries for this indication.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology
* Not have received cytotoxic chemotherapy regimens for metastatic castration-resistant prostate cancer
* Have prostate cancer progression as assessed by the investigator with prostate-specific antigen progression according to Prostate Cancer Working Group 2 criteria
* Have asymptomatic or mildly symptomatic prostate cancer
* Have ongoing androgen deprivation with serum testosterone <50 ng/dL (<2.0 nM)
* Have Eastern Cooperative Oncology Group performance status of <=2
* Laboratory values within protocol-defined parameters
* Adequate liver function according to protocol-defined parameters
* Be able to swallow the study drug whole as a tablet
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* Eligible for another study of abiraterone acetate that is open to enrollment
* Has received abiraterone acetate in the past or was enrolled in Studies COU-AA-301 or COU-AA-302
* Has serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
* Has uncontrolled hypertension (systolic blood pressure >=160 mmHg or diastolic blood pressure >=95 mmHg); individuals with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive therapy
* Has active or symptomatic viral hepatitis or chronic liver disease
* Has a history of pituitary or adrenal dysfunction
* Has clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association Class III or IV heart disease or left ventricular ejection fraction of <50% at baseline
* Has atrial fibrillation or other cardiac arrhythmia
* Has known brain metastasis
* Has had prior cytotoxic chemotherapy or biologic therapy for the treatment of castration-resistant prostate cancer (CRPC)
* Has had prior cytotoxic chemotherapy or biologic therapy for the treatment of CRPC
* Has an active infection or other medical condition that would make prednisone/prednisolone use contraindicated
* Has had other anticancer therapy including cytotoxic, radionucleotide, and immunotherapy
* Has had prior systemic treatment with an azole drug; diethylstilbestrol; PC-SPES; spironolactone; and other preparations such as saw palmetto thought to have endocrine effects on prostate cancer, within 4 weeks of Cycle 1 Day 1
* Is currently enrolled in an investigational drug or device study or has participated in such a study within 30 days of Day 1
* Has a condition or situation which, in the investigator's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with participant's participation in the study
* Has partners of childbearing potential who are not willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator and sponsor during the study and for 13 weeks after last study drug administration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (8):
- Brazil (8):
  - Belo Horizonte
  - Brasília
  - Florianópolis
  - Fortaleza
  - Jaú
  - Porto Alegre
  - Santo André
  - São Paulo

REFERENCES:
- See also: Open-label Study of Abiraterone Acetate plus Prednisone in Asymptomatic or Mildly Symptomatic Subjects with Metastatic Castration-Resistant Prostate Cancer (Early Access Protocol) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR100946&attachmentIdentifier=8deb2b73-eb82-4ba4-8b75-16ff014b1a37&fileName=CR100946_CSR.pdf&versionIdentifier=